CLINICAL TRIAL: NCT03146689
Title: Identifying Treatment Responders to a Topical Non-steroidal Anti-inflammatory Drug (NSAID) or Topical Capsaicin in Painful Knee Osteoarthritis: A Pilot Series of N-of-1 Trials
Brief Title: Ibuprofen Gel or Capsaicin Cream for my Painful Knee Osteoarthritis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Arthritis Research UK Pain Centre (Unknown); Nottingham University Hospitals Charity (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B 10022017
Record Dates: First submitted 2017-05-03; First posted 2017-05-10 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; n-of-1; ibuprofen; capsaicin; NSAID; topical
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Anti-Inflammatory Agents, Non-Steroidal; Ibuprofen; Gels; Capsaicin

STUDY DESIGN:
Intervention Model Description: N-of-1 trial series: several within-individual, randomised, multiple cross-over trials aggregated into a series.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical NSAID and topical capsaicin (Experimental): Within each participant:
  Topical NSAID (A) or capsaicin (B) are taken for a treatment period of four weeks. This is followed by another four week treatment period with the other treatment. These two treatment periods comprise one treatment cycle. The order of treatments within a treatment cycle is determined randomly (AB or BA).
  This treatment cycle is repeated so that all participants undergo a maximum of three topical NSAID treatment periods and three topical capsaicin treatment periods (i.e., three treatment cycles). This is reduced to two cycles if they are found to meet the criteria for response at the interim analysis (after cycle two).
  Interventions: Drug: Topical NSAID; Drug: Topical Capsaicin

INTERVENTIONS:
Drug: Topical NSAID — Applied four times daily
  Other Names: Ibuprofen 5% gel
Drug: Topical Capsaicin — Applied four times daily
  Other Names: Zacin 0.025% cream

SUMMARY:
Despite evidence that topical non-steroidal anti-inflammatory drugs (NSAIDs) and capsaicin are effective in osteoarthritis (OA), it is still unclear why they work for some people but not others. The investigators are undertaking an individual patient data (IPD) meta-analysis to identify responders according to patient characteristics, however, no studies report the presence of synovial hypertrophy or neuropathic-like pain. These two traits are of interest as they may be used to optimise the treatment effects of the two drugs which work via different mechanisms to reduce pain in OA. The investigators are therefore conducting this pilot n-of-1 trial series.

This pilot n-of-1 trial series will investigate whether a person with OA, who has a different balance between inflammatory and neuropathic pain, shows a preference between these mechanistically different treatments. The trial will also be used to offer recommendations on the use of n-of-1 trial series for individualised (precision) medicine in OA.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women who have had ultrasound and radiographic assessments in the Knee Pain in the Community study

  o Premenopausal women will need to be on an acceptable contraceptive method
* Aged 40-95 years
* Knee pain between 4-8 on the NRS
* Knee osteoarthritis - defined as knee pain plus radiographic changes, based on previous questionnaire responses and radiographic findings

  * Knee pain: individuals with knee pain in and around the knee on most days for at least a month.
  * Radiographic changes: definite joint space narrowing and definite osteophytes (each scoring two or more on the Nottingham Line Drawing Atlas) in the tibiofemoral and/or patellofemoral compartments
* Predominantly neuropathic or inflammatory phenotypes based on previous questionnaire responses (not current status)

  * Predominantly neuropathic phenotype: painDETECT Questionnaire (PDQ) > 13 and synovial hypertrophy (SH) <4 mm
  * Predominantly inflammatory phenotype: SH > 4 mm and PDQ < 13
  * If we cannot recruit enough people with the above thresholds, we will base recruitment on the overall distribution of PDQ and SH scores from the population. The third tertile of PDQ and the first tertile of SH for neuropathic and the first tertile of PDQ and the third tertile of SH for inflammatory phenotypes.

Exclusion Criteria:

* Inability to give informed consent
* Daily use of oral NSAIDs for the last two weeks
* Prior use of Ibuprofen gel or Zacin on the affected knee(s)
* Terminal or untreated major mental illness
* Pregnancy or breastfeeding
* Hypersensitivity or allergy to topical NSAIDs, capsaicin, or other ingredients in the preparations. This includes individuals that experience attacks of asthma, urticaria, or acute rhinitis that are precipitated by NSAIDs
* Current treatment for stomach or duodenal ulcers
* Total joint replacement of affected joint
* Renal failure
* Taking anticoagulants

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline knee pain on 0-10 numeric rating scale (NRS) | Baseline and end of each treatment period (i.e., after four weeks of treatment)
  Pain experienced in the most painful knee in the past week will be recorded. The following question will be asked for this purpose: "In the past week, on average, how intense was your knee pain rated on a 0-10 scale, where 0 is 'no pain' and 10 is 'pain as bad as could be'?". The change in pain score between period baseline and period end will be calculated

SECONDARY OUTCOMES:
End-of-cycle treatment preference | At the end of each treatment cycle (i.e., after 4 weeks of NSAID and 4 weeks of capsaicin).
  "Considering only the pain relief experienced in this most recent cycle, which treatment do you feel provided satisfactory pain relief?"
End-of-study overall treatment preference | At study completion - following six treatment periods (24 weeks of treatment, excluding washouts) or 4 treatment periods for responders at the interim analysis (16 weeks of treatment, excluding washouts)
  "Considering all the aspects of the treatment, including its effectiveness and ease of application, which treatment do you prefer?"
Weekly knee pain on 0-10 numeric rating scale (NRS) | At end of week 1, week 2, week 3, and week 4 of each treatment period.
  Pain experienced in the most painful knee in the past week will be recorded. The following question will be asked for this purpose: "In the past week, on average, how intense was your knee pain rated on a 0-10 scale, where 0 is 'no pain' and 10 is 'pain as bad as could be'?".

CONTACTS AND LOCATIONS:
Overall Officials: Weiya Zhang, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Academic Rheumatology, University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Requests for the IPD can be made to the Prof Weiya Zhang. Raw de-identified data may be shared
Supporting Information: Study Protocol
Time Frame: After publication of the study

REFERENCES:
- [Derived] Persson MSM, Stocks J, Sarmanova A, Fernandes G, Walsh DA, Doherty M, Zhang W. Individual responses to topical ibuprofen gel or capsaicin cream for painful knee osteoarthritis: a series of n-of-1 trials. Rheumatology (Oxford). 2021 May 14;60(5):2231-2237. doi: 10.1093/rheumatology/keaa561. PMID 33197270